CLINICAL TRIAL: NCT02697383
Title: Ixazomib (MLN9708) and Dexamethasone in High Risk Smoldering Multiple Myeloma: A Clinical and Correlative Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-294
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma; High Risk Smoldering Multiple Myeloma
Keywords: Ixazomib (MLN9708); Dexamethasone; 15-294
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone

ARMS (1):
- Ixazomib (MLN9708) and Dexamethasone (Experimental): Patients with high risk SMM will be enrolled on the pilot study and treated with 2 drug combination (Cycles 1-12 Ixazomib at 4 mg weekly on days 1, 8 and 15, and dexamethasone on days 1, 8, 15 and 22 of 28 day cycle); the dexamethasone dose will be 40 mg/week the first 4 cycles, thereafter 20 mg/week.
  Interventions: Drug: Ixazomib (MLN9708); Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib (MLN9708)
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to see what effects, good and/or bad, the combination of ixazomib and dexamethasone has on the patient and the smoldering multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Smoldering Multiple Myeloma confirmed by Department of Pathology, based on the International Myeloma Working Group Criteria
* Serum M-protein ≥3 g/dl and/or bone marrow plasma cells ≥10 %,
* Absence of anemia attributed to the plasma cell disorder*: Hemoglobin >10 g/dl or not more than 2g/dL below the lower limit of normal
* Absence of renal failure attributed to the plasma cell disorder*: calculated creatinine clearance (according to Cockcroft-Gault method, MDRD, or CKD-EPI formulae) > 30 mL/min (or alternatively based on standard creatinine level criteria of 2 mg/dl)
* Absence of hypercalcemia attributed to the plasma cell disorder* (: Ca < 10.5 mg/dl or ≤ 2.5 mmol/L
* Absence of lytic bone lesion
* Absence of Clonal bone marrow plasma cell percentage ≥60%
* Absence of Involved: uninvolved serum free light chain ratio ≥100
* Absence >1 focal lesions on MRI studies

  * To be determined based on clinical and laboratory assessment by the primary oncologist
  * "High-risk SMM" per Mayo Clinic or Spanish PETHEMA criteria
  * Measurable disease within the past 4 weeks defined by any one of the following
* Serum monoclonal protein ≥ 1.0 g/dl
* Urine monoclonal protein >200 mg/24 hour
* Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio (reference 0.26-1.65)

  * Age ≥18 years
  * ECOG performance status 0, 1, or 2.
  * Ability to give informed consent.
  * Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count ≥1.0 K/μL
* Platelets ≥ 75 K/μL (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.)
* Hemoglobin > 10 g/dL(transfusions are not permissible)
* Total bilirubin ≤1.5 X institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤ 3.0 X institutional upper limit of normal

  * Female patients who:
* Are postmenopausal for at least 24 months before the Screening visit, OR
* Are surgically sterile, OR
* If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
* Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

  * Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
* Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
* Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Participation in other clinical trials, including those with other investigational agents not included in this trial and throughout the duration of this trial; within at least 5 half-lives of previous therapy for smoldering myeloma at start of this trial.
* Prior therapy for SMM with a proteasome inhibitor.
* Patients with a diagnosis of MM per standard IMWG criteria
* Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Uncontrolled hypertension or diabetes.
* Females patients who are lactating or have a positive serum pregnancy test during the screening period.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Patient has ≥ Grade 1 peripheral neuropathy with pain on clinical examination during the screening period.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before study enrollment, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis.
* Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Psychiatric illness/social situation that would limit compliance with study requirements.
* QTc > 470 milliseconds (msec) on a 12-lead EKG obtained during the Screening period. If a machine reading is above this value, the EKG should be reviewed by a qualified reader and confirmed on a subsequent EKG.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements or GI procedure that could interfere with the oral absorption or tolerance of treatment.
* Major surgery within 14 days prior to enrollment.
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
* Central nervous system involvement (based on clinical assessment).
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* No current anti-myeloma bisphosphonate therapy (however, prior bisphosphonates and/or bisphosphonate therapy due to osteoporosis is allowed).
* Patients with Paget's disease of the bone.
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
best response | up to 12 cycles of treatment (28 day cycle)
  best overall response rate (PR or better) Stringent Complete Response (sCR) Complete Response as defined below plus: Normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence (presence/absence of clonal cells is based on the kappa/ lambda ratio. Complete Response (CR) Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow Very Good Partial Response (VGPR) Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24h Partial Response (PR) ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200mg per 24h. If the serum and urine M-protein are unmeasureable, a ≥50% decrease in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sham Mailankody, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/